CLINICAL TRIAL: NCT05970419
Title: Efficacy Of Non-Invasive High Power Laser Acupuncture Stimulation In Chronic Non-Specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tasnim Mohamed Elfeky, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tasnim Mohamed Elfeky
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Low Back Pain
Keywords: chronic Low Back pain; high-intensity laser therapy; high power laser acupuncture
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High power laser acupuncture group (Experimental): This group will receive high power laser acupuncture (HPLA) +conventional therapy
  Interventions: Other: high power laser acupuncture (HPLA); Other: conventional treatment
- Conventional treatment group (Active Comparator): This group will receive sham laser and The first line of chronic nonspecific low back pain treatment is the conventional treatment.
  Interventions: Other: conventional treatment; Other: Sham laser

INTERVENTIONS:
Other: high power laser acupuncture (HPLA) — High power laser therapy A Zimmer Opton pro, integrated High-power class IV laser device (serial N: 15200013306 & REF: 4682, made in Germany, manufactured by Zimmer Medizin System). It emits radiation in the infrared range to deliver topical heating and raise tissue temperature. The simultaneous application of two wavelengths of laser light (810 and 980nm) provides the user with a huge variety of therapy options. The laser probe - with the small spacer (3.1cm2) , with parameters of 3 watts, 5Hz, 50% duty cycle, 20 joule/ point for 13 seconds with 6.4 j/cm2 . Although a maximum power of 8000 W was reported in two studies, the average power of the lasers used in t
  Arms: High power laser acupuncture group
Other: conventional treatment — Superficial heat (hot packs). Will be applied 10 - 15 minutes. Guideline-endorsed treatment is to stay active, return to normal activity, and to exercise. Different exercise types are used in the treatment of CLBP such as strength and aerobic training on land as well as specific exercises such as motor control exercises (MCE).
  General exercises activating the extensor (paraspinals) and flexor (abdominals) muscle groups will be used.
Other: Sham laser — sham laser (Not active)
  Arms: Conventional treatment group

SUMMARY:
This study will be conducted to answer the following question: Does high power laser acupuncture has any effect on pain, back range of motion, function, quality of life, fatigue and level of satisfaction in chronic nonspecific low back pain patients?

DETAILED DESCRIPTION:
The aims of this study are:

1. To investigate the effect of high power laser acupuncture on pain in chronic nonspecific low back pain patients
2. To investigate the effect of high power laser acupuncture on back range of motion (flexion, extension, side bending and rotation) in chronic nonspecific low back pain patients.
3. To investigate the effect of high power laser acupuncture on function in chronic nonspecific low back pain patients.
4. To investigate the effect of high power laser acupuncture on quality of life in chronic nonspecific low back pain patients.
5. To investigate the effect of high power laser acupuncture on back muscle fatigue in chronic nonspecific low back pain patients.
6. To investigate the effect of high power laser acupuncture on level of satisfaction in chronic nonspecific low back pain patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included in this study will be having all of the following criteria:

1. Age over 18 years of age.
2. Both genders (males and females).
3. Normal BMI ranges between 18.5:24.9 kg/m2.
4. Patients will be referred from an orthopedist with diagnosis of chronic low back pain without underlying pathological causes. The patients with chronic nonspecific low back pain more than 3months. Minimum pain intensity of 30 mm on the visual analogue scale (VAS) for pain, which ranges from 0 to 100 mm.

6) CNSLBP patients will be diagnosed based on the standard criteria, including pain and tenderness on lower back and a negative result for all special tests for lumber neurological examination.

Exclusion Criteria:

1. History of any surgical procedure in the back or the lower extremities.
2. Back pain secondary to known specific pathology (e.g. infection, tumor, osteoporosis, fracture, structural deformity, inflammatory disorder (e.g. ankylosing spondylitis) or cauda equine syndrome).
3. Patient with lumbar instability including spondylolisthesis.
4. Red flags (e.g. fever, unexplained weight loss, progressive weakness, radiation to lower limb, bowel and bladder dysfunction).
5. Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in intensity of pain | at baseline and after 4 weeks of intervention
  By using visual analoge scale (VAS). It is a valid and reliable measure to assess pain intensity level by patients by making a mark determining a decimal number from 0 to 100 (mm) on line with 'no pain' to the left and severe pain could be to the right. The subjects will rate their perception of pain by making a mark on the VAS line. The distance from the left to the mark will be measured and the accuracy will be adjusted to one decimal place.
Assessing the change in Back Range of Motion | at baseline and after 4 weeks of intervention
  By using the Back Range of Motion Instrument (BROM). It is a valid and reliable measure to assess back range of motion (flexion, extension, side bending and rotation) The BROM is uses a patented inclinometer based instrument for measuring lateral side bend in the preferred upright position. The magnetic inclinometer and reference eliminate hip substitution errors. The BROM Basic includes two Universal Inclinometers for measuring flexion and extension of the lumbar spine.
Assessing the change in Quality of Life | at baseline and after 4 weeks of intervention
  By using the short version of the WHO Quality of Life Instrument in Arabic. It will be used to assess quality of life.
  The World Health Organization Quality-of-Life Scale (WHOQOL-BREF) provides a reliable, valid, and brief assessment of quality-of-life. There will be a four-domain score. The four domain scores will denote an individual perception of quality of life in each particular domain. Domains scores are scaled in a positive direction higher score denote higher quality of life. The mean score of items within each domain is used to calculate the domain score. Mean scores are then multiplied by 4 in order to make domain scores comparable with the scores used in the WHOQOL-100.
Assessing the change in endurance of the trunk extensor muscles | at baseline and after 4 weeks of intervention
  By using Biering-Sorensen test. The Sorensen test allows for a rapid, simple, and reproducible evaluation of the isometric endurance of the trunk extensor muscles. It discriminates between healthy individuals and patients with low back pain and may predict the occurrence of low back pain in the near future. The test consists in measuring the amount of time a person can hold the unsupported upper body in a horizontal prone position with the lower body fixed to the examining table.
  The Biering-Sørensen test for measuring back muscle fatigue is valid and provides reliable measures of position-holding time and can discriminate between subjects with and without nonspecific low back pain.
Assessing the change in patient satisfaction | at baseline and after 4 weeks of intervention
  By using The MedRisk Instrument for Measuring Patient Satisfaction (MRPS). A Self-report measures that sample a variety of items provide clinicians with an array of information that may assist in assessing patient satisfaction. The MRPS questionnaire is valid and reliable for measuring patient satisfaction. It has a 2-factor structure: "internal," relating to the patient-therapist interaction, and "external," describing no therapist issues such as admissions and clinic environment.

CONTACTS AND LOCATIONS:
Overall Officials: Tasnim Mohamed, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic faculty of physical therapy cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided